CLINICAL TRIAL: NCT01848483
Title: The Living Well Project: Early Palliative Care and Motivational Interviewing (MI) for Persons With AIDS
Brief Title: Living Well Project for Persons With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Grady Health System (Other)
Responsible Party: Principal Investigator, Marcia McDonnell Holstad, DSN, FNP-BC, Principal Investigator, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00059987; NIH/NINR-1R01NR014054-01 (Other: Other)
Record Dates: First submitted 2013-02-05; First posted 2013-05-07 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Acquired Immunodeficiency Syndrome (AIDS)
Keywords: Early Palliative Care; Motivational Interviewing; Persons Living With Human immunodeficiency virus(HIV); Acquired Immunodeficiency Syndrome (AIDS)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIDS EPC Package plus MI (Experimental): AIDS EPC Package plus MI: AIDS Early Palliative Care (EPC) Package and Motivational Interviewing (MI) At least one early Palliative Care visit plus four weekly MI sessions within a 3 month period of time.
  Interventions: Behavioral: AIDS EPC Package plus MI; Other: Standard of Care (SOC)
- Standard of Care (SOC) (Other): Standard of Care (SOC): Routine Infectious Disease Program HIV-care clinic appointment
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: AIDS EPC Package plus MI — 1. Motivational Interviewing: In MI session #1, the nurse will set the agenda & ask the participant to discuss any adjustments to the AIDS diagnosis. In sessions #2 - 4, the participant will be asked to set the agenda related to current concerns. In sessions #3 & 4, the nurse will also introduce advance care planning.
  2. EPC Package: Participants will be seen by palliative care providers, for approximately 30 minutes each, in the following order: 1) Chaplain: introduces the concept of EPC clinic & conducts a spiritual evaluation/intervention as needed. 2) Social worker: conducts an evaluation/intervention as needed. 3) Psychologist: conducts an evaluation/intervention as needed. 4) Palliative Care Physician: conducts symptom management, medication reconciliation & coordination of care.
  Other Names: Motivational Interviewing; AIDS Early Palliative Care Package
  Arms: AIDS EPC Package plus MI
Other: Standard of Care (SOC) — The routine standard of care provider visit occurs in the following order. The vital signs are taken and the participant sees the nurse to review medications. The provider visits are scheduled for approximately 30 minutes, except for a new patient or patient with complex medical needs. The provider conducts a history to elicit symptoms, health problems, concerns, and a physical exam, then orders labs or immunizations; and referrals to subspecialty clinics. Medications are prescribed or renewed. The patient then receives a follow-up appointment, typically every 3 months for a stable patient. If the patient starts Antiretroviral therapy (ART), an appointment to the nurse educator is required. Typically, the patient will have 1- 2 visits to the nurse educator to begin medications and follow-up for side-effects.

SUMMARY:
The overall goal of this project is to implement and test the efficacy of an enhanced comprehensive multidisciplinary early palliative care (EPC) package that includes four motivational interviewing sessions (MI) for persons diagnosed with AIDS. We posit that the innovative EPC will improve quality of life, clinical and psychosocial outcomes and advance care planning in a cost effective manner and could promote engagement and retention in HIV care. If successful, it could serve as a model of early palliative care for persons with AIDS in the US.

DETAILED DESCRIPTION:
The overall goal of this project is to improve the health and quality of life of persons living with HIV/AIDS (PLWH). To this end, we will implement an innovative model of enhanced early integrative palliative care services (EPC) for persons diagnosed with AIDS. Patients will be recruited from either the inpatient service or outpatient infectious disease program (IDP) at the Grady Health System (GHS) in Atlanta, Georgia. The AIDS EPC Package includes use of motivational interviewing (MI) to facilitate adjustment to disease and advance care planning decision making. The project has three specific aims:

Aim 1. Conduct a research clinical trial (RCT) to examine the efficacy of the AIDS EPC Package intervention vs. standard HIV care (SOC) and compare outcomes at 12 months post baseline. Our hypothesis is that those in the AIDS EPC group will have:

i. Better clinical outcomes: a lower one year mortality, higher proportion who initiate antiretroviral therapy (ART), higher proportion with virologic suppression, higher CD4 gain, fewer opportunistic infections (OI), fewer hospitalizations, lower depression scores, and better symptom management (including cognitive dysfunction).

ii. Better psychosocial outcomes: Better coping skills, higher perceived social support, higher spirituality, higher levels of self-advocacy, lower proportion who report substance use.

iii. Better Quality of Life (QOL) and a higher proportion who report advance care planning activities: named a surrogate; set personal goals regarding life saving measures; and discussed these goals with a surrogate.

SECONDARY OUTCOMES:

Aim 2. Evaluate the cost effectiveness and cost utility of the AIDS EPC Package compared to SOC where the outcomes are valued as survival and quality-adjusted life years (QALYs) respectively.

Aim 3. Promote engagement and retention in HIV care as evidenced by attending a greater proportion of scheduled appointments and reporting higher satisfaction with care compared to SOC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIDS (using current Centers for Disease Control and Prevention criteria)
* Detectable viral load (>1.6 log or > 40 copies per ml)
* Not currently on ART
* Age ≥18 years
* Able to speak and write English
* Able to give and understand consent
* Willing to participate in study activities.

Exclusion Criteria:

* Participants who have a Karnofsky score of 30 or less and are impaired in 5 activities of daily living (ADL) from this list: Bathing, dressing, transferring from bed or chair, walking, eating, toilet use, or grooming
* Those not HIV infected
* Minors under 18 years of age
* Unable to read or understand English
* Cognitive impairment
* Actively psychotic
* Severely depressed/suicidal
* Pose a risk of harm to themselves or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia McDonnell Holstad, phD, Principal Investigator — Emory University
Locations (1):
- Emory University, Nell Hodgson Woodruff School of Nursing, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in June 2014 at Emory University
Groups:
- Standard of Care (SOC): Standard of Care (SOC): Routine Infectious Disease Program HIV-care clinic appointment
  Standard of Care (SOC): The routine standard of care provider visit occurs in the following order. The vital signs are taken and the participant sees the nurse to review medications. The provider visits are scheduled for approximately 30 minutes, except for a new patient or patient with complex medical needs. The provider conducts a history to elicit symptoms, health problems, concerns, and a physical exam, then orders labs or immunizations; and referrals to subspecialty clinics. Medications are prescribed or renewed. The patient then receives a follow-up appointment, typically every 3 months for a stable patient. If the patient starts ART, an appointment to the nurse educator is required. Typically, the patient will have 1- 2 visits to the nurse educator to begin medications and follow-up for side-effects.
Period: Overall Study
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Started | 61 | 60
Completed | 50 | 49
Not Completed | 11 | 11
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Incarceration | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC) | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.2) | 42.3 (10.3) | 42.6 (10.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 46 | 44 | 90
  Female | 13 | 13 | 26
  Transgender | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 58 | 56 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 50 | 106
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121
Sexual Orientation [Count of Participants; unit: Participants]
  Straight/heterosexual | 24 | 28 | 52
  Gay/homosexual | 25 | 21 | 46
  Bisexual | 6 | 6 | 12
  None of de above/unsure | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: Change in Quality of Life (QOL) as measured by the McGill Quality of Life Questionnaire (MQOL) The MQOL has been widely used with persons with a life-threatening illness, including HIV/AIDS. It contains questions about physical wellbeing, physical symptoms, psychological symptoms, existential wellbeing and support in the past 2 days.A total score was computed.Scores range from 0 to 10 with higher scores indicating better perceived quality of life.
Time Frame: Baseline, 3 month post-baseline, 6 month post-baseline, 12 months post-baseline
Population: Only included participants that were able to complete the McGill Quality of Life Questionnaire at each visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Number analyzed (Participants) | 61 | 60
score on a scale
  Baseline | 5.87 (1.62) | 5.17 (1.43)
  3 months post-baseline: number analyzed (Participants) | 50 | 47
  3 months post-baseline | 5.68 (1.73) | 5.06 (1.63)
  6 months post-baseline: number analyzed (Participants) | 51 | 52
  6 months post-baseline | 5.73 (1.90) | 5.09 (1.74)
  12 months post-baseline: number analyzed (Participants) | 50 | 49
  12 months post-baseline | 6.15 (1.73) | 5.30 (1.78)

2. Secondary Outcome: Clinical Indicator: Change in Mortality at 12 Months Post-baseline
Description: Number of deaths at 12 months post baseline
Time Frame: Baseline, up to 12 months post- baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Number analyzed (Participants) | 61 | 60
Participants | 2 | 1

3. Secondary Outcome: Clinical Indicator: Change in Self-report Hospitalizations
Description: Participants completed a survey asking about hospitalizations for HIV related problems and non-HIV related health problems in the past 3 months.Results are expressed in number of participants reporting a hospital stay in the previous 3 months.
Time Frame: Baseline, 3 month post-baseline, 6 month post-baseline, 12 months post-baseline
Population: Participants analyzed in each time point include the ones that were able to complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Number analyzed (Participants) | 61 | 60
Participants
  Baseline HIV related: number analyzed (Participants) | 61 | 59
  Baseline HIV related | 24 | 27
  3 months post-baseline HIV related: number analyzed (Participants) | 49 | 47
  3 months post-baseline HIV related | 11 | 12
  6 months post-baseline HIV related: number analyzed (Participants) | 50 | 53
  6 months post-baseline HIV related | 5 | 10
  12 months post-baseline HIV related: number analyzed (Participants) | 50 | 49
  12 months post-baseline HIV related | 6 | 7
  Baseline non-HIV related: number analyzed (Participants) | 61 | 59
  Baseline non-HIV related | 22 | 23
  3 months post-baseline non-HIV related: number analyzed (Participants) | 50 | 47
  3 months post-baseline non-HIV related | 15 | 15
  6 months post-baseline non-HIV related: number analyzed (Participants) | 49 | 53
  6 months post-baseline non-HIV related | 7 | 17
  12 months post0baseline non-HIV related: number analyzed (Participants) | 49 | 49
  12 months post0baseline non-HIV related | 10 | 12

4. Secondary Outcome: Change in Self-reported Completion of Advanced Care Planning Activities: Health Care Decision Maker
Description: The Advanced Care Planning Questionnaire contained questions about 5 aspects of advanced care planning: 1) advanced care planning decisions made; 2) how well informed a participant feels about medical decision makers and making decisions; 3) how much a person has thought about medical decision making; 4) one's perceived confidence to make medical decisions; 5) one's readiness to make medical decisions. The results focus on decisions made regarding signing papers that name a health care decision maker (yes/no). Results are reported as the number of patients who report "yes".
Time Frame: Baseline, 6 months post-baseline, and 12-months post baseline
Population: Participants analyzed in each time point include the ones that were able to complete the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Number analyzed (Participants) | 61 | 60
Participants
  Baseline | 13 | 12
  6 months post-baseline: number analyzed (Participants) | 51 | 51
  6 months post-baseline | 21 | 11
  12 months post-baseline: number analyzed (Participants) | 50 | 49
  12 months post-baseline | 22 | 16

5. Secondary Outcome: Change in Self-reported Completion of Advanced Care Planning Activities: Living Will
Description: The Advanced Care Planning Questionnaire contained questions about 5 aspects of advanced care planning: 1) advanced care planning decisions made; 2) how well informed a participant feels about medical decision makers and making decisions; 3) how much a person has thought about medical decision making; 4) one's perceived confidence to make medical decisions; 5) one's readiness to make medical decisions. The results focus on decisions made regarding signing papers for either advance directives or living will (yes/no). Results are reported as the number of patients who report "yes".
Time Frame: Baseline, 6 months post-baseline, and 12-months post baseline
Population: Participants analyzed in each time point include the ones that were able to complete the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
Number analyzed (Participants) | 61 | 60
Participants
  Baseline | 12 | 8
  6 months post-baseline: number analyzed (Participants) | 51 | 51
  6 months post-baseline | 14 | 8
  12 months post-baseline: number analyzed (Participants) | 50 | 49
  12 months post-baseline | 19 | 11

ADVERSE EVENTS:
Time Frame: 12 months post baseline
Arm/Group | AIDS EPC Package Plus MI | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 2/61 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT01848483/Prot_SAP_000.pdf